CLINICAL TRIAL: NCT04935021
Title: Clinical Study Protocol of Transthyroxine Protein Amyloidosis Cardiomyopathy and Its Gene Carriers
Brief Title: Clinical Study of ATTR-CM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0132
Record Dates: First submitted 2021-06-20; First posted 2021-06-22 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Transthyroxine Amyloidosis Cardiomyopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATTR-CM (Experimental): Patients or Gene carrier
  Interventions: Drug: ATTR-CM

INTERVENTIONS:
Drug: ATTR-CM — Current treatment

SUMMARY:
In this study, patients with ATTR-CM or gene carriers were selected to study the diagnosis and treatment, and long-term follow-up was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patients and gene carriers of ATTR-CM confirmed in the Second Affiliated Hospital of Zhejiang University School of Medicine, regardless of gender, age 18-90 years old;
* Patients who have the ability to understand the test and can cooperate with investigators

Exclusion Criteria:

* Patients who unable to understand or unwilling to fill in informed consent forms or follow visitors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2031-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of cardiovascular death, myocardial infarction, and stroke | 10 year
  Primary Outcome

CONTACTS AND LOCATIONS:
Locations (1):
- xiaohong University PAN, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided